CLINICAL TRIAL: NCT05914103
Title: The Application of Enhanced Recovery After Surgery (ERAS) for Cardiovascular Surgery in the Correction of Complex Congenital Heart Disease: a Stepped Wedge Cluster Randomized Trial
Brief Title: The Application of Enhanced Recovery After Surgery (ERAS) for Cardiovascular Surgery in the Correction of Complex Congenital Heart Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Fuwai Yunnan Cardiovascular Hospital (Other); Beijing Anzhen Hospital (Other); The Second People's Hospital of GuangDong Province (Other); Shanghai Children's Medical Center (Other)
Responsible Party: Principal Investigator, Yan Fuxia, principal investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-1969
Record Dates: First submitted 2023-05-17; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Complex Congenital Heart Disease; Enhanced Recovery After Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Procedure: ERAS
- Control (No Intervention)

INTERVENTIONS:
Procedure: ERAS — The primary endpoint is the rate of composite outcomes. The composite outcomes include the major adverse cardiac events (MACE), major postoperative pulmonary complication (PPCs), and acute kidney injury (AKI)
  Arms: Intervention

SUMMARY:
This study is a multicenter, stepwise design, cluster randomized controlled trial. Random sequence is generated by computer, and each center enters the intervention expectation (Phase I) in random order to implement ERAS strategy. If it does not enter the intervention expectation (Phase C) center, clinical diagnosis and treatment will be completed according to the traditional scheme.

Among children, patients aged 28 to 6 who underwent cardiac surgery were included in the ERAS strategy intervention plan, which mainly includes preoperative education, preoperative comfort for the patient, preoperative oral sugary beverage, continuous infusion of dexmedetomidine, multimodal analgesia, blood protection strategies, prevention of postoperative nausea and vomiting, intraoperative insulation, early tracheal extubation and intubation, and targeted liquid therapy. The traditional plan group follows the current clinical diagnosis and treatment routine. By comparing the differences in the incidence of major postoperative outcomes (MACE events, major pulmonary complications, and acute kidney injury) between the intervention group and the non intervention group, as well as comparing other adverse events (including but not limited to pneumonia, massive bleeding, postoperative arrhythmia, incision infection, postoperative nausea, vomiting, and delirium), all cause secondary intubation, and all cause secondary surgery between the two groups, and recording hospitalization time, ICU stay time The removal time of tracheal intubation and drainage tube, the pain score during hospitalization, the total amount of opioid drug use (converted to the same dose of morphine), hospitalization expenses, and family satisfaction scores were recorded to explore whether the ERAS regimen can reduce the incidence of major postoperative adverse events, improve patient prognosis, and accelerate postoperative recovery compared to traditional regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 28 days to 6 years
* Patients awaiting elective cardiac surgery with cardiopulmonary bypass (CPB).

Exclusion Criteria:

* The risk adjustment for congenital heart surgery (RACHS) is above class 5
* Patients with cardiac assist device, mechanical ventilation or the history of asphyxia
* Patients with pulmonary disease, including respiratory tract infections and asthma
* Patients with severe liver or renal dysfunction, including severe acute or chronic renal dysfunction need renal replacement therapy, and acute or chronic liver failure need artificial liver therapy
* Fetal malformation includes polysplenia syndrome, Asplenia Syndrome, Down syndrome, DiGeoge syndrome, Marfan syndrome, trachea-bronchus stricture, diabetes, nervous functioning disorders, genital system malformations, imperforate anus, and Williams syndrome
* Current enrollment in another clinical trial
* Guardian's refusal or low adherence

Ages: 28 Days to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3030 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
composite outcomes | during hospitalization, an average of 1 week, assessed up to 30 days
  The composite outcomes include the major adverse cardiac events (MACE), major postoperative pulmonary complication (PPCs), and acute kidney injury (AKI)

SECONDARY OUTCOMES:
length of hospital stay | From the date of admission until the date of discharging, assessed up to 30 days
  From the date of admission until the date of discharging
the duration of intensive care unit (ICU) stay | Time from ICU admission to ICU discharge, assessed up to 30 days
  Time from ICU admission to ICU discharge
time to extubation | The time from the end of operation to the removal of tracheal intubation, assessed up to 30 days
  The time from the end of operation to the removal of tracheal intubation
time to drainage removal | The time from the end of operation to the removal of drainage tube, assessed up to 30 days
  The time from the end of operation to the removal of drainage tube
the rate of other complications | during hospitalization, an average of 1 week, assessed up to 30 days
  The rate of other complications include delium, pneumonia, pneumothorax, hematorrhea and so on
the rate of reintubation for any cause | during hospitalization, an average of 1 week, assessed up to 30 days
  The rate of reintubation for any cause
cumulative opioid dosage | during hospitalization, an average of 1 week, assessed up to 30 days
  Total perioperative consumption of opioid analgesics
overall medical costs | during hospitalization, an average of 1 week, assessed up to 30 days
  Total cost of patients during hospitalization
Satisfaction score | the day before discharge, assessed up to 30 days
  A satisfaction rating using a 0-10 number scale (0=unsatisfactory, 10=satisfactory)
the cumulative incidence of death from any cause within 30 days and 1 year | within 30 days and 1 year
  the cumulative incidence of death from any cause within 30 days and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yan, Principal Investigator — Fuxia hospital
Locations (2):
- China (2):
  - Fuwai hospital, Beijing, Beijing Municipality
  - Fuwai hospital, China, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dou D, Jia Y, Yuan S, Wang Y, Li Y, Wang H, Ding J, Wu X, Bie D, Liu Q, An R, Yan H, Yan F. The protocol of Enhanced Recovery After Cardiac Surgery (ERACS) in congenital heart disease: a stepped wedge cluster randomized trial. BMC Pediatr. 2024 Jan 5;24(1):22. doi: 10.1186/s12887-023-04422-2. PMID 38183047